CLINICAL TRIAL: NCT00320775
Title: An Exploratory Study of the Safety, Tolerability and Biological Effect of Intravitreal Administration of VEGF Trap in Patients With Neovascular Age-Related Macular Degeneration
Brief Title: Safety and Tolerability Study of Intravitreal VEGF-Trap Administration in Patients With Neovascular AMD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VGFT-OD-0502
Record Dates: First submitted 2006-04-28; First posted 2006-05-03 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Macular Degeneration
Keywords: Neovascular Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part A (Experimental): Part A: An open label study in which six successive cohorts of 3-6 patients each with neovascular AMD will receive a single intravitreal (ITV) injection of 0.05, 0.15, 0.5, 1.0, 2.0, or 4.0 mg of VEGF Trap into the study eye. The total volume of each injection will be 100 μL. Enrollment in new dose levels will not begin until all patients in the preceding dose level have completed Visit 5 (Day 15).
  Interventions: Drug: VEGF Trap
- Part B (Active Comparator): Part B: A controlled, prospective, randomized, double-masked study in which up to 30 subjects meeting eligibility criteria will be randomly assigned in a 1:1 ratio to receive a single ITV injection of2.0 mg/eye VEGF Trap (or the MTD if reached prior to 2.0 mg) followed by 1 sham injection six weeks later, or an initial dose of 0.3 mg pegaptanib sodium into the study eye, followed by a second dose six weeks later. Enrollment into Part B will begin 2 weeks after the last subject to receive the 2.0 mg/eye dose in Part A has been observed for 15 days and it has been determined that the safety profile of VEGF Trap at this dose level is adequate to support expansion of dosing at this dose level. The dose of pegaptanib sodium will be 0.3 mg, according to the package insert.
  Interventions: Drug: VEGF Trap
- Part C (Active Comparator): Part C: A controlled, prospective, randomized, double-masked study in which approximately 30 subjects meeting eligibility criteria will be randomly assigned in a 1:1 ratio to receive up to two ITV injections of either 0.15 or 4.0 mg/eye VEGF Trap. Initiation of Part C is contingent upon the 4.0 mg dose being adequately tolerated in Part A.
  Interventions: Drug: VEGF Trap

INTERVENTIONS:
Drug: VEGF Trap — Part A: Six successive cohorts of 3-6 patients each with neovascular AMD will receive a single intravitreal (ITV) injection of 0.05, 0.15, 0.5, 1.0, 2.0, or 4.0 mg of VEGF Trap into the study eye.
  Part B: Up to 30 subjects will be randomly assigned in a 1:1 ratio to receive a single of 2.0 mg/eye VEGF Trap followed by 1 sham injection six weeks later, or an initial dose of 0.3 mg pegaptanib sodium into the study eye, followed by a second dose six weeks later.
  Part C: Approximately 30 subjects will be randomly assigned in a 1:1 ratio to receive up to two ITV injections of either 0.15 or 4.0 mg/eye VEGF Trap.
  After completion of Visit 8 (Day 57), patients from all parts of the study, may be eligible to continue in Open-label Extension and will receive 4.0 mg of VEGF Trap.
  Other Names: Aflibercept

SUMMARY:
The purpose of this trial is to assess the ocular and systemic safety and tolerability of a single intravitreal injection of VEGF Trap in patients with subfoveal choroidal neovascularization (CNV) due to AMD.

DETAILED DESCRIPTION:
This study consists of three parts, Part A, Part B and Part C. Part A is a dose escalation. Part B was terminated early. The (one) subject who received Macugen is not discussed in this website. Part C had subjects receive one of two doses of VEGF Trap (0.15 mg or 4.0 mg).

This is the first study in which human subjects received intravitreal injections of VEGF Trap in a study eye.

ELIGIBILITY:
Inclusion Criteria:

* Subfoveal CNV secondary to AMD.
* Central retinal/lesion thickness ≥ 250µm as measured by optical coherence tomography (OCT).
* ETDRS best-corrected visual acuity of:

  * 20/40 (73 letters) or worse
* Clear ocular media and clear lens(es) to permit good quality stereoscopic fundus photography.

Exclusion Criteria:

* Prior treatment with VEGF Trap, bevacizumab or ranibizumab.
* Any investigational agent within 12 weeks of Visit 2 (Day 1).
* Presence of other causes of CNV.
* Active ocular infection.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2005-06; Primary Completion 2008-06 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability, bioeffect | From baseline to Day 43

SECONDARY OUTCOMES:
The effect of VEGF Trap administration on excess central retinal/lesion thickness | From baseline to Day 43
Best-corrected Early Treatment of Diabetic Retinopathy Study (ETDRS) visual acuity | From baseline to Day 43
Extent of CNV leakage | From baseline to Day 43
Anti-VEGF Trap antibodies in the systemic circulation | From baseline to Day 43
Plasma levels of VEGF Trap | From baseliene to Day 43

CONTACTS AND LOCATIONS:
Overall Officials: Avner Ingerman, MD, Study Director — Regeneron Pharmaceuticals
Locations (8):
- United States (8):
  - Retina Centers, PC, Tuscon, Arizona
  - Loma Linda University Health Care, Loma Linda, California
  - University of Chicago, Chicago, Illinois
  - Johns Hopkins Hospital School of Medicine, Baltimore, Maryland
  - Charlotte Eye, Ear, Nose & Throat Asssociates, Charlotte, North Carolina
  - Dean A. McGee Eye Institute, Oklahoma City, Oklahoma
  - Retina Diagnostic and Treatment Assoc., LLC, Philadelphia, Pennsylvania
  - Retina-Vitreous Associates, P.C., Nashville, Tennessee

REFERENCES:
- [Result] Nguyen QD, Campochiaro PA, Shah SM, Browning DJ, Hudson HL, Sonkin PL, Hariprasad SM, Kaiser PK, Slakter J, Haller JA, Do DV, Mieler W, Chu K, Ingerman A, Vitti R, Berliner AJ, Cedarbaum J; Clear-It 1 Investigators. Evaluation of very high- and very low-dose intravitreal aflibercept in patients with neovascular age-related macular degeneration. J Ocul Pharmacol Ther. 2012 Dec;28(6):581-8. doi: 10.1089/jop.2011.0261. Epub 2012 Jul 9. PMID 22775078
- [Result] Do DV, Schmidt-Erfurth U, Gonzalez VH, Gordon CM, Tolentino M, Berliner AJ, Vitti R, Ruckert R, Sandbrink R, Stein D, Yang K, Beckmann K, Heier JS. The DA VINCI Study: phase 2 primary results of VEGF Trap-Eye in patients with diabetic macular edema. Ophthalmology. 2011 Sep;118(9):1819-26. doi: 10.1016/j.ophtha.2011.02.018. Epub 2011 May 5. PMID 21546089
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/22775078
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/21546089